CLINICAL TRIAL: NCT07129460
Title: Efficacy and Safety of Berberine for Gastric Intestinal Metaplasia: a Prospective, Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Efficacy and Safety of Berberine for Gastric Intestinal Metaplasia
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Yongquan Shi, Professor, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY20252248-F-1
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Gastric Intestinal Metaplasia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Berberine group (Experimental): Patients in the Berberine group will receive oral Berberine hydrochloride at a dosage of 300 mg two times daily for 6 months
  Interventions: Drug: Berberine hydrochloride
- The placebo group (Placebo Comparator): Patients in the placebo group will receive oral placebo at a dosage of 300 mg two times daily for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Berberine hydrochloride — Subjects will be instructed to take three tablets (300mg) of Berberine hydrochloride two times daily, and visit the hospital every 4 weeks for evaluation of the subjective symptoms and to receive a new supply of medication.
  Arms: The Berberine group
Drug: Placebo — Subjects will be instructed to take three tablets (300mg) of placebo two times daily, and visit the hospital every 4 weeks for evaluation of the subjective symptoms and to receive a new supply of medication.
  Arms: The placebo group

SUMMARY:
The goal of this clinical trial is to investigate the efficacy of Berberine in treating gastric intestinal metaplasia in Helicobacter pylori-negative adults. It will also learn about the safety of Berberine. The main questions it aims to answer are:

Does Berberine promote the regression of IM in individuals without Helicobacter pylori infection? What medical problems do participants experience when taking Berberine? Researchers will compare Berberine to a placebo (a look-alike substance that contains no drug) to see if uBerberine is effective in treating gastric intestinal metaplasia.

Participants will:

TakeBerberine or a placebo every day for 6 months. Visit the clinic once every 4 weeks for checkups and tests.

ELIGIBILITY:
Inclusion Criteria:

* patients aged from 18 to 75 years old.
* patients with OLGIM stage Ⅱ-Ⅳ diagnosed by upper gastrointestinal endoscopy and histopathological examination within the last 3 months.
* patients without Helicobacter pylori infection, including patients who had successful Helicobacter pylori eradication before enrollment.

Exclusion Criteria:

* a history of regular use (defined as at least once per week) of non-steroidal anti-inflammatory drugs (NSAIDs) and/or statins/or Metformin.
* a history of stomach surgery (including endoscopic submucosal dissection and endoscopic mucosal resection) or previously diagnosed malignant tumor.
* a history of heart failure, renal failure, liver cirrhosis or chronic hepatic failure; patients with contraindications or allergies to the drugs in this study.
* breastfeeding or pregnancy.
* a history of substance abuse or alcohol abuse within the past one year.
* patients with severe mental illness.
* refusal to undergo drug treatment.
* refusal to sign informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
The regression rate of gastric intestinal metaplasia based on OLGIM stage in different groups. | From enrollment to the end of treatment at 6 months
  Regression was defined as a OLGIM stage decreased at least one grade.
The progression rate of gastric intestinal metaplasia based on OLGIM stage in different groups. | From enrollment to the end of treatment at 6 months
  Progression was defined as a OLGIM stage increased at least one grade.

SECONDARY OUTCOMES:
The regression rate of gastric atrophy based on OLGA stage in different groups. | From enrollment to the end of treatment at 6 months
  Regression was defined as a OLGA stage decreased at least one grade.
The progression rate of gastric atrophy based on OLGA stage in different groups. | From enrollment to the end of treatment at 6 months
  Progression was defined as a OLGA stage increased at least one grade.

IPD SHARING:
Plan to Share IPD: No